CLINICAL TRIAL: NCT01148667
Title: Interaction of Orally Administered Lactobacillus Rhamnosus GG With Skin and Gut Microbiota and Humoral Immunity in Infants With Atopic Dermatitis
Brief Title: Lactobacillus Rhamnosus GG: Interaction With Human Microbiota and Immunity
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Turku University Hospital (Other Government)
Collaborators: Academy of Finland (Other); Mead Johnson Nutrition (Industry)
Responsible Party: Prof. Erika Isolauri, University of Turku
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 12/2006 1 531
Record Dates: First submitted 2010-06-21; First posted 2010-06-22 (Estimated); Last update posted 2010-06-22 (Estimated); Status verified 2010-06

CONDITIONS: Gut Microbiota; Skin Microbiota; Humoral Immune Responses; Severity of Atopic Dermatitis
Keywords: atopic dermatitis; barrier function; gut; probiotics; skin
MeSH Terms: conditions — Dermatitis, Atopic

STUDY DESIGN:
Who Masked: Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Infants drink formula added with LGG (Active Comparator): Infants have been randomized (1:1) to get casein hydrolysate with or without LGG
  Interventions: Dietary Supplement: Casein hydrolysate added with LGG
- Infants drink casein hydrolysate without LGG (Placebo Comparator): Infants get extensively hydrolysed casein formula
  Interventions: Dietary Supplement: Infants drink casein hydrolysate without LGG

INTERVENTIONS:
Dietary Supplement: Casein hydrolysate added with LGG — Infants drink extensively hydrolysed casein formula supplemented with LGG (ATCC 53103) 5.0 x 10 7 cfu/g to achieve a daily intake of 3.4 10 9 cfu.
  Arms: Infants drink formula added with LGG
Dietary Supplement: Infants drink casein hydrolysate without LGG — Infants drink extensively hydrolysed casein formula without added LGG
  Arms: Infants drink casein hydrolysate without LGG

SUMMARY:
Hypothesis: Probiotics have been used as novel adjunct therapeutic approach in atopic dermatitis. In addition to balancing the gut microecology and promoting host immune defences, specific probiotics might further aid in controlling the microbial colonization of the skin, thereby reducing proneness to secondary infections which typically cause sustained symptoms.

Thirty-nine infants with atopic dermatitis,randomized for a three-month-period in a double-blind design to receive extensively hydrolysed casein formula (NutramigenR, Mead-Johnson, USA) supplemented with (n=19) or without (n=20) Lactobacillus rhamnosus GG (ATCC 53103) 5.0 x 107 cfu/g to achieve a daily intake of 3.4 x 109 cfu.

Sampling (blood and faecal samples, cotton swab from the skin) and clinical examination of the infant, including SCORAD assessment to determine the severity of atopic dermatitis, at each study visit (at entry and one month and three months thereafter).

ELIGIBILITY:
Inclusion Criteria:

* clinical diagnosis of atopic dermatitis
* age 4 we - 18 mo

Exclusion Criteria:

* skin infection or severe infection at the time of enrollment

Ages: 4 Weeks to 18 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Actual)
Dates: Start 2007-03; Primary Completion 2008-07 (Actual); Study Completion 2008-07 (Actual)

PRIMARY OUTCOMES:
severity of atopic dermatitis | March 2007 - July 2008
  Severity of atopic dermatitis of the study infants will be assessed by SCORAD index

SECONDARY OUTCOMES:
Maturation of humoral immune responses | March 2007 - July 2008
  Determination of proportions of immunoglobulin secreting cells among peripheral blood mononuclear cells was carried out by ELISPOT assay. The proportions of CD 19+ memory B cells was carried out by flow cytometry

CONTACTS AND LOCATIONS:
Locations (1):
- Turku University Central Hospital, Turku, Finland

REFERENCES:
- [Derived] Nermes M, Kantele JM, Atosuo TJ, Salminen S, Isolauri E. Interaction of orally administered Lactobacillus rhamnosus GG with skin and gut microbiota and humoral immunity in infants with atopic dermatitis. Clin Exp Allergy. 2011 Mar;41(3):370-7. doi: 10.1111/j.1365-2222.2010.03657.x. Epub 2010 Dec 1. PMID 21121981